CLINICAL TRIAL: NCT00140842
Title: Neuroendocrine Modulation of Metabolic Effects in Overweight Adolescents
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Chief, Pediatric Endocrinology, Massachusetts General Hospital
Other Study IDs: 2004-P-002191
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: Obesity, adolescent, ghrelin, growth hormone, cortisol
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese girls: The inclusion criteria will be girls 12-18 years of age. According to the Centers for Disease Control and Prevention, the definition of obesity is a BMI higher than the 95th percentile for age and sex, and that of overweight is a BMI between the 85th and 95th percentiles. Cases will be defined as having a body mass index (BMI) greater than the 95th percentile for age according to the 2000 Centers for Disease Control and Prevention growth charts.
- Normal-weight girls

SUMMARY:
This study will examine hormonal differences in ghrelin and growth hormone in obese and normal weight adolescents and their relationship to body composition and insulin resistance. The study will also investigate the effect of the macronutrient composition of a meal on postprandial ghrelin levels and whether ghrelin responses will predict the degree of hunger and caloric intake at a subsequent meal.

DETAILED DESCRIPTION:
Obesity is an epidemic that is striking people at younger ages than ever before. Obesity is associated with changes in the secretory patterns of several hormones including ghrelin, growth hormone (GH), and insulin, which have not been examined in the adolescent age group. Ghrelin, a primarily gastric hormone, increases appetite and is a GH secretagogue. This study will compare the alteration in secretion of ghrelin and GH in overweight and normal weight adolescent girls through frequent blood sampling and GH stimulation testing with growth hormone releasing hormone and arginine. The relationship between these hormones and insulin resistance, measured by 1H-nuclear magnetic resonance spectroscopy, and body composition, measured by dual energy x-ray absorptiometry and magnetic resonance imaging, will be investigated. This study will also determine the postprandial ghrelin response to test meals that vary by the type of predominant macronutrient, which may predict the degree of hunger and amount of intake at a subsequent meal. Understanding obesity-related changes in ghrelin and GH and their relationship to body composition, insulin resistance, and appetite will help in the development of strategies to reduce complications of obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Girls 12-18 years of age
2. Obese subjects: BMI higher than the 95th percentile for age and sex
3. Normal-weight controls: BMI from the 15th to the 85th percentiles for age and sex

Exclusion Criteria:

1. History of disorders other than obesity that may affect growth hormone, ghrelin, cortisol, or insulin secretion such as eating disorder, diabetes mellitus, hypertension, thyroid disease, Cushing's syndrome, liver disease, renal failure, or an excess or deficiency of GH or cortisol
2. Medications that could affect glucose and lipid levels or the secretion of growth hormone, ghrelin, insulin, or cortisol such as rhGH, glucocorticoids, and birth control pills
3. Pregnancy
4. Smoking or substance abuse
5. Active dieting
6. Surgical procedures for obesity
7. Dietary restrictions such as bread, dairy, peanut, aspartame, or meat products used in the study
8. Metal implants, including intracranial surgical clips or pacemakers

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese and normal-weight girls between 12-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Misra M, Tsai PM, Mendes N, Miller KK, Klibanski A. Increased carbohydrate induced ghrelin secretion in obese vs. normal-weight adolescent girls. Obesity (Silver Spring). 2009 Sep;17(9):1689-95. doi: 10.1038/oby.2009.86. Epub 2009 Mar 26. PMID 19325538
- [Result] Misra M, Bredella MA, Tsai P, Mendes N, Miller KK, Klibanski A. Lower growth hormone and higher cortisol are associated with greater visceral adiposity, intramyocellular lipids, and insulin resistance in overweight girls. Am J Physiol Endocrinol Metab. 2008 Aug;295(2):E385-92. doi: 10.1152/ajpendo.00052.2008. Epub 2008 Jun 10. PMID 18544645
- [Result] Russell M, Bredella M, Tsai P, Mendes N, Miller KK, Klibanski A, Misra M. Relative growth hormone deficiency and cortisol excess are associated with increased cardiovascular risk markers in obese adolescent girls. J Clin Endocrinol Metab. 2009 Aug;94(8):2864-71. doi: 10.1210/jc.2009-0380. Epub 2009 May 12. PMID 19435823
- [Result] Russell M, Mendes N, Miller KK, Rosen CJ, Lee H, Klibanski A, Misra M. Visceral fat is a negative predictor of bone density measures in obese adolescent girls. J Clin Endocrinol Metab. 2010 Mar;95(3):1247-55. doi: 10.1210/jc.2009-1475. Epub 2010 Jan 15. PMID 20080853
- See also: Click here for more information about this study: Neuroendocrine Modulation of Metabolic Effects in Overweight Adolescents — http://www.massgeneral.org/an/studies_healthy.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 obese and 30 normal-weight adolescents (12-18 yr old) were screened for study eligibility.15 obese adolescents completed the study visit. These subjects were matched for race, ethnicity, and bone age to normal-weight adolescents from the pool of screened subjects.
Groups:
- Normal-weight Girls: Normal weight girls 12-18 years old
- Obese Girls: Obese adolescents between 12-18 years old.
Period: Overall Study
Arm/Group | Normal-weight Girls | Obese Girls
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal-weight Girls: Normal-weight girls were required to have a BMI between the 15th-85th percentiles
- Obese Girls: Obese girls were required to have a BMI above the 95th percentile
- Total: Total of all reporting groups
Arm/Group | Normal-weight Girls | Obese Girls | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (1.7) | 14.0 (1.9) | 14.9 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Growth Hormone (GH) on the GH Stimulation Test
Description: Peak growth hormone (GH) on the GH stimulation test is a measure of the adequacy of GH secretion.
Time Frame: Baseline
Population: This was a cross-sectional study to compare differences in growth hormone (GH) secretory status in relation to body composition in obese versus normal-weight girls. This was a pilot study and the analysis was performed using a Student t-test to compare means across groups
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Normal-weight Girls | Obese Girls
Number analyzed (Participants) | 15 | 15
ng/ml | 40.1 (16.1) [0 to 100] | 25.2 (21.8)
Statistical Analysis 1: Comparison: Normal-weight Girls vs Obese Girls; The null hypothesis was that there is no difference between the groups for peak growth hormone on the growth hormone stimulation test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 15, Standard Deviation 16

2. Secondary Outcome: Visceral Adipose Tissue
Description: Visceral adipose tissue was measured using magnetic resonance imaging at the level of the fourth lumbar vertebra (L4)
Time Frame: Baseline
Population: The analysis was completed on the 30 participants as per protocol
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Normal-weight Girls | Obese Girls
Number analyzed (Participants) | 15 | 15
grams | 19 (7.5) [0 to 100] | 42.7 (17.0) [0 to 100]
Statistical Analysis 1: Comparison: Normal-weight Girls vs Obese Girls; The null hypothesis is that there is no difference between the groups for visceral adipose tissue; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 23.7, Standard Deviation 12

ADVERSE EVENTS:
Arm/Group | Normal-weight Girls | Obese Girls
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Limited number of participants-pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No